CLINICAL TRIAL: NCT07263191
Title: A Multicenter, Prospective Observational Study to Evaluate Treatment Patterns and Safety in Patients With Bipolar Disorder Taking Olanzapine
Brief Title: A Study of Olanzapine in Participants With Bipolar Disorder.
Status: Recruiting | Type: Observational
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: BR-OLZ-OS-401
Record Dates: First submitted 2025-11-23; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Bipolar Disorder
Keywords: Olanzapine; Observation study; Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Olanzapine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Olanzapine — As this is a non-interventional study designed to collect data as part of routine clinical practice, the selection and dosage of medication, treatment period, and whether or not to change it are all based on the clinician's judgment.

SUMMARY:
This study aimed to identify treatment patterns in patients with bipolar disorder receiving olanzapine according to demographic and clinical characteristics and to evaluate the effectiveness of education on weight gain, a side effect of olanzapine, in preventing weight gain.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have signed the informed consent after receiving information about the purpose and method of this study.
* Patients diagnosed with bipolar disorder and scheduled to receive olanzapine.
* Patients who understand the contents of the survey and can answer the questions directly.

Exclusion Criteria:

* Female patients who are pregnant, have childbearing potential, or are breastfeeding.
* Has received an investigational product within 12 weeks from the study enrollment or has plans to participate in another clinical trial during the participation of this study.
* Other subjects who are considered inappropriate to participate in this study by the judgment of the investigator.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with bipolar disorder who require olanzapine administration
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2025-10-30 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Treatment pattern | Baseline, 8weeks, 12weeks
  Frequency and percentage of the therapeutic class of bipolar disorder agents administered within 8 weeks prior to baseline will be presented based on the patients' demographic factors and clinical characteristics. Furthermore, frequency and percentage of the therapeutic class patterns of bipolar disorder agents administered after baseline will be presented

SECONDARY OUTCOMES:
Change From Baseline in Young Mania Rating Scale (YMRS) Score at 8 Weeks and 12Weeks. | Baseline, 8weeks, 12weeks
  The YMRS scoring system ranges from 0 (no symptoms) to 4 or 8 (severe symptoms)
Change From Baseline in Patient Health Questionnaire-9 (PHQ-9) Score at 8 Weeks and 12Weeks. | Baseline, 8weeks, 12weeks
  The PHQ-9 scoring system ranges from 0 to 27, with higher scores indicating more severe depression. Each item is scored on a scale from 0 to 3
Change From Baseline in Clinical Global Impression Scale-Severity (CGI-S) Score at 8 Weeks and 12Weeks. | Baseline, 8weeks, 12weeks
  The CGI is rated on a 7-point scale, with the severity of illness scale using a range of responses from 0 (not assessed) through to 7 (amongst the most severely ill patients).
Clinical Global Impression Scale-Improvement (CGI-I) scores at 8 and 12 weeks after drug administration | Baseline, 8weeks, 12weeks
  The CGI is rated on a 7-point scale, with the severity of illness scale using a range of responses from 0 (not assessed) through to 7 (amongst the most severely ill patients).
Adverse events | Up to 27months

CONTACTS AND LOCATIONS:
Locations (1):
- CHA Bundang Medical Center, Seongnam, South Korea

IPD SHARING:
Plan to Share IPD: No